CLINICAL TRIAL: NCT01237119
Title: 48-week Phase II, Randomised, Double Blinded Placebo Controlled Multicentre Trial on Liraglutide's Safety, Efficacy and Action on Liver Histology and Metabolism in Overweight Patients With NASH +/- Type II Diabetes
Brief Title: Liraglutide Efficacy and Action in Non-Alcoholic Steatohepatitis
Acronym: LEAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Wellcome Trust (Other); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HE2013; ISRCTN85774727 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Experimental): A once-daily glucagon-like peptide 1 (GLP-1) analogue. Currently has regulation approval for use in type 2 diabetics (ref: guidelines)
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): Liraglutide-Placebo manufactured by Novo Nordisk.
  Interventions: Other: Liraglutide-placebo

INTERVENTIONS:
Drug: Liraglutide — 1.8 mg once daily, subcutaneous injection
  Other Names: Victoza
  Arms: Liraglutide
Other: Liraglutide-placebo — 1.8 mg once-daily, subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate whether 48 weeks treatment with once-daily injections of liraglutide improves liver disease (liver fat, inflammation and scarring) and related metabolic parameters in overweight patients with nonalcoholic steatohepatitis, enough to warrant further investigation.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is responsible for an increasing prevalence of liver disease and is becoming the commonest cause of liver disease in the western world. NAFLD is recognised to be the hepatic manifestation of the metabolic syndrome, which is a cluster of metabolic abnormalities characterised by abdominal obesity, insulin resistance, impaired glucose metabolism, hypertension and dyslipidaemia. In its mildest form there is an accumulation of fat in the liver (steatosis) without any liver damage, however in many cases it progresses to non-alcoholic steatohepatitis (NASH), and cirrhosis.

Current treatment options for NASH are limited in efficacy, necessitating the development of more effective options. New agents such as Glucagon-like Peptide-1 (GLP-1) agonists that improve diabetic control and facilitate weight loss have been suggested as therapies in NASH.

No published studies to date have assessed the impact of the GLP-1 agonist, Liraglutide, on liver histology and metabolism in obese patients with NASH. This study hypothesises that treatment with liraglutide will result in a significant improvement in histological disease activity in overweight patients with NASH, in the presence or absence of Type 2 Diabetes (T2DM)

ELIGIBILITY:
Inclusion Criteria:

* NASH on liver biopsy (within 6 months of screening visit).
* NAFLD Activity Score (NAS) ≥ 3, comprising of a minimum of 1 point from each of the individual steatosis, lobular inflammation and hepatocyte ballooning scores
* Body Mass Index (BMI) ≥ 25 at randomisation
* Type 2 Diabetes Mellitus/impaired glucose tolerance or normal glucose tolerance

Exclusion Criteria (brief):

* Insulin dependent diabetes
* Glycosylated Haemoglobin (HbA1c) > 9.0%
* treatment with dipeptidyl peptidase 4 (DPP-IV) inhibitors, Glucagon-like Peptides (GLP) 1 analogues, thiazolidinediones (TZDs)
* Past Medical History of Acute (or chronic) pancreatitis/pancreatic carcinoma, weight loss surgery, liver transplantation, Medullary thyroid cancer, hepatocellular carcinoma (HCC), Multiple Endocrine Neoplasia (MEN) syndrome, malignancy (within last 3 years, exception of treated skin malignancy)
* Other liver aetiologies (i.e. drug-induced, viral hepatitis, autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, haemochromatosis, alpha 1 anti-trypsin deficiency, Wilsons disease)
* concomitant or recent use of orlistat, prednisolone,
* Refusal or lacks capacity to give informed consent to participate in the trial
* Participation in any clinical trial of an investigational therapy or agent within 3 months of randomisation
* Patient (or carer) deemed not competent at using the correct site and technique for subcutaneous injection of the trial treatment (containing dummy drug on practice) at visit 2
* NAS<3
* Child's B or C cirrhosis
* Abnormal clinical examination of thyroid (i.e. unexplained goitre or palpable nodules)
* Liver enzymes > 10 x upper limit of normal
* Average alcohol consumption per week > 21 units (210g) male, >14 units (140g) female within the last 5 years.
* >5% weight loss since the diagnostic liver biopsy was obtained.
* Recent or concomitant use of steroids (oral), methotrexate, amiodarone, Orlistat
* Addition or significant change (as judged by the chief investigator) in dose of the following drugs; Angiotensin converting enzymes (ACE)-inhibitors, Angiotensin receptor blockers (ARBs) and/or Multi-vitamins (containing Vitamin E)
* Known positivity for antibody to Human Immunodeficiency virus (HIV)
* Serum creatinine > 150 μmol/L or currently being treated with renal replacement therapy
* Past medical history of multiple drug allergies (defined as anaphylactoid drug reactions in >2 drug groups)
* Presence of any acute/chronic infections or illness that at the discretion of the chief investigator might compromise the patient's health and safety in the trial
* Pregnancy or breastfeeding
* Women, of child-bearing age, who are not willing to practise effective contraception (i.e. barrier, oral contraceptive pill, implanon or history hysterectomy) for the 48 week duration of the trial and for one-month after the last administration of the drug.
* Men, sexually active with women of child-bearing age, who are not willing to practise effective contraception for the 48 week duration of the trial and for one-month after the last administration of the drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Liver Histological improvement | 48 weeks

SECONDARY OUTCOMES:
NAFLD Activity Score | 48 weeks
  Also including:
  Fibrosis panel, Liver Function Tests (LFTs), cytokeratin-18 (CK-18) Glycaemic control, Fibroscan, Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Philip N Newsome, FRCPE PhD, Principal Investigator — Centre for liver research, University of Birmingham
Locations (1):
- NIHR BRU Centre for liver research, Queens Elizabeth University Hospital Birmingham, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Background] Armstrong MJ, Barton D, Gaunt P, Hull D, Guo K, Stocken D, Gough SC, Tomlinson JW, Brown RM, Hubscher SG, Newsome PN; LEAN trial team. Liraglutide efficacy and action in non-alcoholic steatohepatitis (LEAN): study protocol for a phase II multicentre, double-blinded, randomised, controlled trial. BMJ Open. 2013 Nov 4;3(11):e003995. doi: 10.1136/bmjopen-2013-003995. PMID 24189085
- [Result] Armstrong MJ, Gaunt P, Aithal GP, Barton D, Hull D, Parker R, Hazlehurst JM, Guo K; LEAN trial team; Abouda G, Aldersley MA, Stocken D, Gough SC, Tomlinson JW, Brown RM, Hubscher SG, Newsome PN. Liraglutide safety and efficacy in patients with non-alcoholic steatohepatitis (LEAN): a multicentre, double-blind, randomised, placebo-controlled phase 2 study. Lancet. 2016 Feb 13;387(10019):679-690. doi: 10.1016/S0140-6736(15)00803-X. Epub 2015 Nov 20. PMID 26608256
- [Result] Armstrong MJ, Hull D, Guo K, Barton D, Hazlehurst JM, Gathercole LL, Nasiri M, Yu J, Gough SC, Newsome PN, Tomlinson JW. Glucagon-like peptide 1 decreases lipotoxicity in non-alcoholic steatohepatitis. J Hepatol. 2016 Feb;64(2):399-408. doi: 10.1016/j.jhep.2015.08.038. Epub 2015 Sep 21. PMID 26394161